CLINICAL TRIAL: NCT05133375
Title: Comparison of Hemodynamic Changes of Tracheal Intubation With McCoy and Macintosh Laryngoscopes
Brief Title: Hemodynamic Changes of Tracheal Intubation With McCoy and Macintosh Laryngoscopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Jhelum (Other)
Responsible Party: Principal Investigator, M. Awais Qarni, Anesthesiologist, CMH Jhelum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11112021
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Hemodynamic Rebound
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): Macintosh laryngoscope was used for endotracheal intubation.
  Interventions: Procedure: Tracheal Intubation
- GROUP B (Experimental): McCoy laryngoscope was used for endotracheal intubation.
  Interventions: Procedure: Tracheal Intubation

INTERVENTIONS:
Procedure: Tracheal Intubation — Before reporting to Operation theatre, a detailed pre anesthesia assessment was done in all patients, all necessary laboratory investigations were collected. On OT table pulse and systolic blood pressure was checked by non-invasive method. 18G cannula was passed and ECG was attached. A pillow was placed under the head to obtain classical sniffing position for intubation. All the patients were pre medicated with injection midazolam 0.08mg/kg, injection nalbuphine 0.1 mg/kg, injection dexamethasone 0.08mg/kg and injection metoclopramide 0.1 mg/kg. Pre oxygenation was done with 100% oxygen for 3 mins. Induction was done with injection propofol2 mg/kg, muscle relaxation achieved with injection atracurium 0.5mg/kg. Laryngoscopy was started after 3 minutes by a qualified anesthetist. Pulse and systolic blood pressure was recorded by non-invasive measures before laryngoscopy and at 30 seconds, 2 and 3 minutes after intubation.

SUMMARY:
A total of 272 patients were randomly allocated into two groups, Patients in group A were treated with Macintosh laryngoscope and in groups B with McCoy laryngoscope was used for endotracheal intubation. Pulse and systolic blood pressure was recorded by non-invasive measures before laryngoscopy and at 30 seconds, 2 and 3minutes after intubation. All this information was recorded on a Pro forma.

DETAILED DESCRIPTION:
After taking approval from hospital ethical committee, 272 patients who reported to Operation Theatre of CMH, Jhelum were selected for the study. Informed consent was obtained and patient demographic information (name, age, contact) was recorded. Patients were randomly divided in two equal groups by using lottery method. GROUP A: Where Macintosh laryngoscope was used for endotracheal intubation. GROUP B: Where McCoy laryngoscope was used for endotracheal intubation.

Before reporting to Operation theatre a detailed pre anesthesia assessment was done in all patients, all necessary laboratory investigations were collected. On OT table pulse and systolic blood pressure was checked by non-invasive method. 18G cannula was passed and ECG was attached. A pillow was placed under the head to obtain classical sniffing position for intubation. All the patients were pre medicated with injection midazolam 0.08mg/kg, injection nalbuphine 0.1 mg/kg, injection dexamethasone 0.08mg/kg and injection metoclopramide 0.1 mg/kg. Pre oxygenation was done with 100% oxygen for 3 mins. Induction was done with injection propofol2 mg/kg, muscle relaxation achieved with injection atracurium 0.5mg/kg. Laryngoscopy was started after 3 minutes by a qualified anesthetist. Pulse and systolic blood pressure was recorded by non-invasive measures before laryngoscopy and at 30 seconds, 2 and 3minutes after intubation. All this information was recorded on a Proforma.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female
* Age between 18 to 70
* ASA I and II males and females.
* Malampatti I and II.
* Hemodynamically stable, no known ischemic heart disease and no history of hypertension.
* Nil per oral for at least 6 hours.

Exclusion Criteria:

* Non consenting patient.
* ASA III, IV or V patient.
* Malampati III or IV.
* Cervical instability
* Thyromental distance of less than 6cm, inter incisor distance of less than 3cm.
* Known case of hypertension and ischemic heart disease.
* Pregnant female.
* Body mass index of more than 30.
* Patients of oropharyngeal surgery.
* Unable to Intubate in less than 1 minute.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Effect on the pulse of intubation with Macintosh and McCoy laryngoscope | After Laryngoscopy, pulse was recorded by non-invasive measures before laryngoscopy and at 30 seconds, 2 and 3 minutes after intubation.
  To measure hemodynamic changes (i.e. pulse) of intubation with Macintosh and McCoy laryngoscope
Effect on the systolic blood pressure of intubation with Macintosh and McCoy laryngoscope | After Laryngoscopy, systolic blood pressure was recorded by non-invasive measures before laryngoscopy and at 30 seconds, 2 and 3 minutes after intubation
  To measure hemodynamic changes (i.e. systolic blood pressure) of intubation with Macintosh and McCoy

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Awais Qarni, Principal Investigator — Anesthesiologist
Locations (1):
- CMH, Jhelum, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Overall results will be shared.